CLINICAL TRIAL: NCT05738967
Title: Transdiagnostic Behavioral Therapy for Anxiety and Depression in Autistic Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Texas Higher Education Coordinating Board (Other Government)
Responsible Party: Principal Investigator, Eric A Storch, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-52639
Record Dates: First submitted 2023-02-08; First posted 2023-02-22 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Depression; Emotional Disorder; Autism
Keywords: Cognitive behavioral therapy; CBT; exposure therapy; behavioral activation
MeSH Terms: conditions — Anxiety Disorders; Depression; Autistic Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transdiagnostic cognitive behavioral therapy (Experimental)
  Interventions: Behavioral: Transdiagnostic cognitive behavioral therapy (CBT)
- Treatment as usual (Active Comparator)
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Transdiagnostic cognitive behavioral therapy (CBT) — Adolescent-caregiver dyads will will participate in CBT focused on exposure therapy and behavioral activation. It will also include flexible incorporation of emotion-focused coping and adaptations for autism.
  Other Names: CBT
  Arms: Transdiagnostic cognitive behavioral therapy
Behavioral: Treatment as usual — Adolescent-caregiver dyads will participate in coordinated referrals to the community. They may receive psychotherapy and/or initiate or change current psychiatric medication (if applicable).
  Other Names: TAU
  Arms: Treatment as usual

SUMMARY:
This study tests the effectiveness of a transdiagnostic cognitive behavioral therapy for autistic youth with anxiety and/or depression.

DETAILED DESCRIPTION:
About 1 in 54 adolescents are estimated to be on the autism spectrum, with over half suffering from anxiety or depressive disorders. These disorders contribute to suicidality, family stress, social impairments, and difficulties transitioning to adulthood among autistic youth. Given the frequency of anxiety and depressive disorders among autistic adolescents and the increased risk of impairment, developing effective treatments for anxiety and depression tailored to this population is a top priority.

Transdiagnostic cognitive behavioral therapy (CBT) for other populations, including typically developing adolescents, may confer broader benefits than disorder-specific CBT and facilitate broader dissemination and implementation. However, there has been little research conducted on transdiagnostic treatments among autistic adolescents. Thus, this study proposes to address this gap by testing transdiagnostic CBT for autistic adolescents with anxiety and depression.

The study involves two phases: 1) a pilot intervention; and 2) a randomized controlled trial.

The pilot intervention will involve 12 adolescent-caregiver dyads to further refine the treatment model and its assessment measures. The randomized trial will involve 100 adolescent-caregiver dyads to further evaluate the clinical efficacy of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Child is between the ages of 12-17 at consent/assent.
* The child meets criteria for autism spectrum disorder using evidence-based assessment approaches (e.g., Autism Diagnostic Observation Schedule-Second Edition; Childhood Autism Rating Scale-Second Edition).
* The child meets criteria for clinically significant anxiety and/or depression symptoms based on elevated scores on the Pediatric Anxiety Rating Scale modified for Autism Spectrum Disorder (>11) and/or the Children's Depression Rating Scale-Revised (>39).
* Anxiety/depressive disorder is the primary presenting problem as determined by administration of the Mini International Neuropsychiatric Interview
* One parent/guardian is able and willing to participate.
* The parent/guardian is 18 years or older.
* Both parent and child can read and/or understand English.
* Both parent and child reside in Texas.

Exclusion Criteria:

* The child has a diagnosis of psychotic disorder and/or conduct disorder.
* The child has severe suicidal/homicidal ideation and/or self-injury requiring immediate intervention and/or a higher level of care.
* The child has limited verbal communication abilities.
* The child is receiving concurrent psychotherapy for anxiety/depression.
* The child has initiated psychotropic medications within 12 weeks of assessments (or 4 weeks for stimulants/benzodiazepines) or during therapy, and/or has changed dosage of psychotropic medication within 6 weeks of assessment (or 2 weeks for stimulants/benzodiazepines) or during therapy.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Revised Children's Anxiety and Depression Scale - Parent-Report | 7 days
  Parent-rated child anxiety and depression severity. It is a 47-item scale. Each item is scored on a 0 ("never") to 3 ("always") scale (higher scores correspond to greater severity), yielding a total between 0 and 141.
Clinical Global Impression - Improvement | 7 days
  Clinician-rated child internalizing symptom improvement since initial rating. A single item is scored 0-6 (0 = very much worse; 6 = very much improved).
Clinical Global Impression - Severity of Illness | 7 days
  Clinician-rated child internalizing symptom overall severity. A single item is scored 0-6 (0 = no illness; 6 = extremely severe symptoms).

SECONDARY OUTCOMES:
Revised Children's Anxiety and Depression Scale - Self-Report | 7 days
  Child rated anxiety and depression severity. It is a 47-item scale. Each item is scored on a 0 ("never") to 3 ("always") scale (higher scores correspond to greater severity), yielding a total between 0 and 141.
Pediatric Anxiety Rating Scale modified for Autism | 7 days
  Clinician-rated child anxiety severity. The rating scale first includes a checklist of common anxiety symptoms that are rated as present/absent and is followed by a severity rating scale with five Likert scale items. Each severity item is scored on a 0 to 5 scale, (higher scores correspond to greater severity), yielding a total between 0 and 30.
Children's Depression Rating Scale, Revised | 7 days
  Clinician-rated child depression severity. It is a 17-item scale, with items ranging from 1 to 5 or 1 to 7 (higher scores correspond to greater severity), yielding a total between 17 and 113.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Psychiatry Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan on publishing the study description, protocol/procedures, and raw data on an OSF website once primary results are published.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available once the primary results are published in a peer-reviewed journal

REFERENCES:
- [Background] Weersing VR, Brent DA, Rozenman MS, Gonzalez A, Jeffreys M, Dickerson JF, Lynch FL, Porta G, Iyengar S. Brief Behavioral Therapy for Pediatric Anxiety and Depression in Primary Care: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Jun 1;74(6):571-578. doi: 10.1001/jamapsychiatry.2017.0429. PMID 28423145
- [Background] van Steensel FJ, Bogels SM, Perrin S. Anxiety disorders in children and adolescents with autistic spectrum disorders: a meta-analysis. Clin Child Fam Psychol Rev. 2011 Sep;14(3):302-17. doi: 10.1007/s10567-011-0097-0. PMID 21735077
- [Background] Hudson CC, Hall L, Harkness KL. Prevalence of Depressive Disorders in Individuals with Autism Spectrum Disorder: a Meta-Analysis. J Abnorm Child Psychol. 2019 Jan;47(1):165-175. doi: 10.1007/s10802-018-0402-1. PMID 29497980
- [Background] Chu BC, Crocco ST, Esseling P, Areizaga MJ, Lindner AM, Skriner LC. Transdiagnostic group behavioral activation and exposure therapy for youth anxiety and depression: Initial randomized controlled trial. Behav Res Ther. 2016 Jan;76:65-75. doi: 10.1016/j.brat.2015.11.005. Epub 2015 Nov 19. PMID 26655958
- [Background] Uljarevic M, Hedley D, Rose-Foley K, Magiati I, Cai RY, Dissanayake C, Richdale A, Trollor J. Anxiety and Depression from Adolescence to Old Age in Autism Spectrum Disorder. J Autism Dev Disord. 2020 Sep;50(9):3155-3165. doi: 10.1007/s10803-019-04084-z. PMID 31190198
- [Background] Wood JJ, Kendall PC, Wood KS, Kerns CM, Seltzer M, Small BJ, Lewin AB, Storch EA. Cognitive Behavioral Treatments for Anxiety in Children With Autism Spectrum Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2020 May 1;77(5):474-483. doi: 10.1001/jamapsychiatry.2019.4160. PMID 31755906